CLINICAL TRIAL: NCT00793091
Title: A Phase 2, Randomized, Placebo-Controlled, Double-Masked, Multicenter Safety and Efficacy Study of C-KAD Ophthalmic Solution in Patients With Loss of Visual Acuity Due to Age-Related Cataract
Brief Title: Safety and Efficacy Study of an Ophthalmic Solution in Patients With Age-Related Cataract
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chakshu Research, Inc. (Industry)
Responsible Party: Watiri Kamau-Kelley, Manager, Clinical & Regulatory Affairs, Chakshu Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CK-0109
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: C-KAD Ophthalmic Solution
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C-KAD Ophthalmic Solution — 4 drops applied daily for 120 days
  Arms: 1
Drug: Placebo — 4 drops applied daily for 120 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of C-KAD Ophthalmic Solution in improving visual acuity relative to placebo in patients with age-related cataract

ELIGIBILITY:
Inclusion Criteria:

* Presence of age-related cataract in the study eye
* Best-corrected visual acuity of 20/25 to 20/50 in the study eye

Exclusion Criteria:

* Any other clinical condition in the eye that may compromise vision
* Presence or History of Glaucoma
* Presence or history of diabetes
* Use of eyedrops
* Use of steroids

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity by ETDRS | 120 Days

CONTACTS AND LOCATIONS:
Overall Officials: Ira Wong, MD, Study Director — Chakshu Research, Inc.
Locations (4):
- United States (4):
  - Pacific Eye Specialists, San Francisco, California
  - Hunkeler Eye Institute, Overland Park, Kansas
  - Minnesota Eye Consultants, PA, Minneapolis, Minnesota
  - Charlotte Eye, Ear, Nose & Throat Associates, Charlotte, North Carolina